CLINICAL TRIAL: NCT05907356
Title: Comparison of Sciatic Nerve Slider Technique in Different Positions in Patients With Low Back Pain Associated With Sciatica: Randomized Control Trial
Brief Title: Effect of Sciatic Nerve Slider Technique in Different Positions in Low Back Pain Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: European University of Lefke (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BAYEK022.06
Record Dates: First submitted 2023-05-28; First posted 2023-06-18 (Actual); Last update posted 2024-08-27 (Actual); Status verified 2024-08

CONDITIONS: Low Back Pain; Sciatica
Keywords: low back pain; Neuromobilization; Sciatic nerve Slider technique; Positions
MeSH Terms: conditions — Low Back Pain; Sciatica | interventions — Supine Position

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Study Group One (Experimental): sciatic nerve slider technique in a slump lying position in combination with Conventional physiotherapy
  Interventions: Other: sciatic nerve slider technique in slump lying position; Other: Conventional physiotherapy
- Study Group Two (Experimental): sciatic nerve slider technique in a supine position in combination with Conventional physiotherapy
  Interventions: Other: sciatic nerve slider technique in supine position; Other: Conventional physiotherapy
- Control Group (Experimental): Conventional physiotherapy alone
  Interventions: Other: Conventional physiotherapy

INTERVENTIONS:
Other: sciatic nerve slider technique in slump lying position — The patient will be sitting at the edge of the couch with the posterior aspect of the knee at the edge, the thighs parallel to each other, and flexion at the thoracic and lumbar spines (slouch position). The therapist will be standing at the bedside of the patient with a proximal arm over the patient's shoulder and one hand guiding the neck movements of the patient and the other hand guiding the knee movements, passively performing cervical neck flexion with knee flexion (stretching the nerve proximally and relaxing at the distal end) and then moving into cervical extension with knee extension. Provide five sets in every session: the first: 10 repetitions, the second: 15 repetitions, the third: 20 repetitions, the fourth: 25 repetitions; and the fifth: 30 repetitions. The end position is held for 5 seconds, and the rest between sets is 1-2 minutes
  Arms: Study Group One
Other: sciatic nerve slider technique in supine position — .The patient will be in a supine position. The therapist will hold the patient's limb passively and then move the hip into flexion with the ankle in plantar flexion and the knee in extension, stretching the nerve at the hip and relaxing at the ankle, Then reversing the movement with the hip into extension, maintaining the knee in extension and the ankle in dorsiflexion, relaxing the nerve at the hip and stretching at the ankle. Provide five sets in every session; the first: 10 repetitions, the second: 15 repetitions, the third: 20 repetitions, the fourth: 25 repetitions, and the fifth: 30 repetitions. The end position is held for 5 seconds, and the rest between sets is 1-2 minutes.
  Arms: Study Group Two
Other: Conventional physiotherapy — The patient will receive conventional physiotherapy, which includes: a moist hot pack, TENS, and back strengthening exercises (as a home program).

SUMMARY:
Neural mobilization is a technique that plays an important role in repairing the neural tissue's ability to respond to stress or tension by triggering the reconstruction of normal physiological functioning, pain reduction, and functional improvement. The study aims to examine the effect of the sciatic nerve slider technique in different positions and which of the most common positions is more effective in the application of neural mobilization in low back pain with sciatica.

DETAILED DESCRIPTION:
Low back pain (LBP) is one of the most common musculoskeletal disorders, accounting for a significant portion of disability. It's a severe healthcare burden that has large societal costs, according to estimates, LBP can affect anywhere between 22% and 65% of people within a year. Additionally, back pain-related absences from work result in prolonged periods of sick leave, which has an adverse effect on workplace productivity.

Sciatica is the name given to a collection of symptoms caused by compression and irritation of the sciatic nerve, including pain, numbness, muscular weakness, and difficulty moving or controlling the legs. The lower back, buttocks, and multiple dermatomes of the leg and foot are typically where symptoms appear. Sciatica can be caused by a disc bulge or herniation, lumbar canal stenosis, spondylolisthesis, trauma, piriformis syndrome, or spinal tumors. It affects women more than men and people who lead sedentary lifestyles more than active ones. It might arise quickly or gradually with physical activity, and it is usually unilateral.

The slider and tensioner are two distinct types of neural mobilization procedures. There are clinical improvements and positive therapeutic benefits after treatment with different neural mobilization techniques, but the slider technique is safer, involves less stretching and strain of the nerves, and has a more significant effect than the tensioner technique.

ELIGIBILITY:
Inclusion Criteria:

* Age range between 40 - 65 years,
* Both genders,
* Diagnosed by magnetic resonance imaging to confirm disc lesion,
* LBP with radicular pain for more than 12 weeks up to 1 year with no acute episodes in the last 4 weeks, and a numeric pain rating score (NPRS) greater than 4/10.
* Positive SLR test with reproduction of neurological symptoms.

Exclusion Criteria:

* Sciatica due to other pathologies (e.g. lumbar canal stenosis or piriformis syndrome),
* Having any physiotherapy before 6 months.
* History of spinal surgery
* Vertebral fracture or trauma,
* Negative SLR test,
* pregnant.

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2023-04-01 (Actual); Primary Completion 2023-11-20 (Actual); Study Completion 2023-12-25 (Actual)

PRIMARY OUTCOMES:
Numeric Pain Rating Scale (NPRS) | 4 weeks
  A numeric pain rating scale (NPRS) will be used to evaluate pain intensity. The scale has a length of 10 cm and a range of 0-10, Here, a score of zero (zero) denotes the absence of pain, a score of one to three (1-3) denotes mild pain, a score of three to five (moderate pain), and a score of six to ten (severe pain)
Oswestry Disability Index (ODI) | 4 weeks
  The disability caused by low back pain will be measured via the Arabic version of the Oswestry Disability Index. The patient will fill out the questionnaire in about 5 minutes, and then the therapist will score it in about 1 minute. The patient marks the most relevant answer for each question as accurately as they can. The scoring system employs a numerical scale from 0 to 5, with the first possible answer being 0 and the last possible answer being 5. The maximum possible score for each section is 5. All the scores will be added together and divided by the total number of possible points to calculate the total score
Modified Schober test | 4 weeks
  Lumbar flexion flexibility will be measured by the modified Schober test. The patient will be standing, and the examiner will mark the L5 spinous process by drawing a horizontal line across the patient's back. A second line is marked 10 cm above the first line. The patient is then instructed to flex forward as if attempting to touch his/her toes, and the examiner remeasures the distance between two lines with the patient fully flexed. The difference between the measurements in the erect and flexion positions indicates the outcome of the lumbar flexion.
Hand-held dynamometry | 4 weeks
  The hand-held dynamometer has good to excellent reliability and validity for most measures of muscle strength, it portable device that is an appropriate and convenient method to assess lower limb muscle strength. to Assessment of isometric muscle strength and power will be performed with the participants in three positions (seated, supine, and prone); hip flexors, knee extensors, and knee flexors were assessed in a seated position; ankle plantar flexors, ankle dorsiflexors, hip abductors, and hip adductors in a supine position; hip extensors in a prone position
Flexible ruler | 4 weeks
  The lumbar lordosis will be measured by a flexible ruler. It is commonly used to measure the degree of spinal curvature of the lumbar lordosis in the sagittal plane. It is a safe, easy-to-use, and inexpensive tool.

CONTACTS AND LOCATIONS:
Overall Officials: Beliz Belgen Kaygisiz, PT, PhD, Principal Investigator — European University of Lefke
Locations (1):
- Princess Alia Governmental Hospital, Hebron, West Bank, Palestinian Territories

IPD SHARING:
Plan to Share IPD: No